CLINICAL TRIAL: NCT01514812
Title: A Double Blind, Randomized, Two Period Crossover Study To Determine The Effect of Multiple Doses of 120 MG Modified Release Formulation of YM150 on the Steady State Pharmacokinetics of Digoxin in Healthy Subjects
Brief Title: A Study to Investigate the Effect of YM150 on the Plasma Concentration of Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 150-CL-007; 2004-004930-15 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Healthy; Pharmacokinetic of Digoxin
Keywords: YM150; digoxin; drug-drug interaction; Plasma concentration; darexaban; Pharmacokinetics of digoxin
MeSH Terms: interventions — darexaban; Digoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- YM150-placebo sequence group (Experimental): YM150+digoxin; Washout; Placebo+digoxin
  Interventions: Drug: YM150; Drug: placebo; Drug: digoxin
- placebo-YM150 sequence group (Experimental): Placebo+digoxin; Washout; YM150+digoxin
  Interventions: Drug: YM150; Drug: placebo; Drug: digoxin

INTERVENTIONS:
Drug: YM150 — oral - modified release formulation of YM150
  Other Names: darexaban
Drug: placebo — oral
Drug: digoxin — oral

SUMMARY:
This study is to evaluate the effect of YM150 on the plasma concentration of digoxin in healthy subjects.

DETAILED DESCRIPTION:
The study will be of a double blind, randomized, two period crossover design. Two treatments, digoxin in combination with YM150, and digoxin in combination with placebo, will be evaluated. Each subject will receive both treatments in random order. Placebo will be used to maintain the blind. Males and females will be equally divided over the treatment orders.

Subjects will be dosed with digoxin and either YM150 or placebo for 8 days to reach steady state. In the second period the subjects will receive digoxin and the alternate treatment. There will be a washout period of at least 10 days between the consecutive treatments. In both study periods the subjects will be admitted the day prior to study drug administration (Day 0). The subjects will be discharged on Day 10. Approximately one week after the last discharge, the subjects will return to the unit for a post study visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as judged by the investigator or sub-investigator based on the results of physical examinations and all tests
* Body weight: male: ≥60 kg, <100 kg; female: ≥45.0 kg, <80.0 kg
* BMI (at screening): ≥18.0, <30.0

Exclusion Criteria:

* Female subjects of child-bearing potential, not practicing adequate methods to prevent pregnancies, like abstinence or double barrier methods
* Known or suspected hypersensitivity / allergy to FXa inhibitors, digoxin, or heart glycosides in general or the constituents of the formulations used
* History of and/or any sign or symptom indicating current abnormal hemostasis or blood dyscrasia, including but not limited to neutropenia, thrombocytopenia, thrombocytopathy, thromboasthenia, hemophilia, Von Willebrand's disease, and vascular purpura, bleeding gums, or frequent nose bleeding
* Family history of congenital vascular malformation (e.g. Marfan's Syndrome) and/or bleeding disorder (e.g. hemophilia, Von Willebrand's disease, Christmas disease)
* PT or aPTT at the screening visit outside the normal range
* History of peptic ulcer or of any other organic lesion susceptible to bleed
* Any surgical intervention (including tooth extraction) or trauma within the last 3 months preceding the initiation of the study
* Any clinically significant history of upper gastrointestinal symptoms (such as nausea, vomiting, abdominal discomfort or upset, or heartburn) in the 4 weeks prior to admission to the Research Unit
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic
* Any of the liver function tests (ALAT, ASAT, LDH and γ-GT) above the upper limit of normal range (ULN)
* Any clinically significant abnormality following the investigator's review of the prestudy physical examination, ECG and clinical laboratory tests
* Abnormal pulse rate and blood pressure measurements at the pre-study visit as follows: Pulse rate <40 or >90 bpm; systolic blood pressure <95 or >160 mmHg; diastolic blood pressure <40 or >95 mmHg (measurements taken after subject has been resting in supine position for 5 min)
* Regular use of any prescribed or OTC (over-the-counter) drugs (including natural and herbal remedies and especially those with P-gp inhibiting activity, like St. John's worth) in the four weeks prior to admission to the Research Unit OR any use of such drugs (including natural and herbal remedies) as well as vitamins in the two weeks prior to admission to the Research Unit
* Donation of blood or blood products within 3 months prior to admission to the Research Unit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-02; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Cmax of digoxin assessed by its plasma concentration change | for 24 hour after the last dose of each period
AUC of digoxin assessed by its plasma concentration change | for 24 hour after the last dose of each period

SECONDARY OUTCOMES:
Changes in the blood coaggregation indexes such as PT(INR), aPTT and FXa | before dosing and 5hr after dosing on days 4 and 8 and 24h and 48h after the last dose
Safety assessed by the incidence of adverse events, vital signs, 12-lead ECG and labo-tests | for 10 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Paris, France

REFERENCES:
- [Derived] Kadokura T, Groenendaal D, Heeringa M, Mol R, Verheggen F, Garcia-Hernandez A, Onkels H. Darexaban (YM150), an oral direct factor Xa inhibitor, has no effect on the pharmacokinetics of digoxin. Eur J Drug Metab Pharmacokinet. 2014 Mar;39(1):1-9. doi: 10.1007/s13318-013-0141-1. Epub 2013 Jun 11. PMID 23754514